CLINICAL TRIAL: NCT00320242
Title: An Open Label Study to Assess the Efficacy of Visual Cues in the Form of the Laser Cane or the U-Step Walker With Laser Accessory in Parkinson's Disease Patients Who Experience Freezing of Gait.
Brief Title: Laser Light Cues for Gait Freezing in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, David K. Simon, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006P000085
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; laser cane; freezing of gait; visual cues
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 mo baseline (Active Comparator): 1 mo baseline before visual cue: Cane or walker, no laserlight visual cue x 1 mo; + laserlight visual cue for 2nd mo
  Interventions: Device: 1 mo baseline before visual cue
- 2 month baseline (No Intervention): Cane or walker, no laserlight visual cue x 2 mo, + laserlight visual cue for 3rd mo

INTERVENTIONS:
Device: 1 mo baseline before visual cue — Laser Cane with Laser Accessory and/or U-Step Walker with Laser Accessory
  Other Names: U-Step Walking Stabilizer
  Arms: 1 mo baseline

SUMMARY:
The purpose of this study is to gather data to see if the Laser Cane and/or U-Step Walker with laser accessory is more effective in aiding with gait freezing than a regular cane/U-Step Walker in patients who have idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
Freezing of gait is a significant clinical problem in Parkinson's disease (PD). It interferes with daily functioning and quality of life and often results in falls that potentially can inflict serious injury. In recent years, much more attention has been focused on the clinical characteristics of gait freezing, the severity of falls that can result, and the use of visual cues as a possible treatment in order to understand the implications of episodic freezing. Few clinical studies have been done to confirm the clinical observations to date. The laser cane is a device that has been used and prescribed in movement disorder centers as the only form of treatment for freezing of gait. Although it has been shown to be effective in many cases, there is no published data to support what has been observed in the clinic. The proposed study seeks to clarify unanswered questions regarding the laser cane and its efficacy in aiding with episodic gait freezing and falls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or a designated proxy have given informed consent
* Subject has been diagnosed with idiopathic Parkinson's disease
* Subject is ambulatory. If a wheelchair is used part-time, it must be used for less than 50% of the time
* Positive assessment for Questionnaire Used to Identify Freezing of Gait in PD Patients at subject's best "on"

Exclusion Criteria:

* Presence of atypical features suggestive of MSA, PSP, ataxia, unexplained or prominent pyramidal signs, and/or autonomic dysfunction
* Subjects who are non-ambulatory more than 50% of the time
* Subjects who have had a history of syncope in the 6 months prior to screening
* Subjects with moderate or advanced dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K Simon, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Neurological Institute of New York at Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No
Some individual participant data was included in the publication. There is no plan to share additional individual participant data.

REFERENCES:
- [Background] Donovan S, Lim C, Diaz N, Browner N, Rose P, Sudarsky LR, Tarsy D, Fahn S, Simon DK. Laserlight cues for gait freezing in Parkinson's disease: an open-label study. Parkinsonism Relat Disord. 2011 May;17(4):240-5. doi: 10.1016/j.parkreldis.2010.08.010. Epub 2010 Sep 3. PMID 20817535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited by movement disorders specialists seen during their clinic visits at either of the 2 participating hospitals
Pre-assignment Details: 6 of the original 32 subjects who had agreed to participate in the study dropped out before any exposure to the laserlight visual cue. Therefore, data are presented only for the 26 subjects who actually participated in the study, includign exposure to this laserlight visual cue.
Groups:
- 1 mo Baseline Before Visual Cue: 1 mo baseline using the cane/walker without the laserlight visual cue, followed by additional time using the visual cue
- 2 Month Baseline Before Visual Cue: 2 month baseline using the laserlight visual cue, followed by 1 additional month using the laserlight visual cue. This group served as an active comparator control for comparison with Group 1during the 2nd month, when group 1 did use the visual cue but group 2 continued without the visual cue.
Period: Overall Study
Arm/Group | 1 mo Baseline Before Visual Cue | 2 Month Baseline Before Visual Cue
Started | 16 | 16
Completed | 14 | 12
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: 32 subjects initially signed the consent form, but 6 dropped out prior to any exposure to the laserlight visual cue. Therefore, data in this study are included for the 26 subjects who entered the study and were eventually exposed to the laserlight visual cue.
Groups:
- All Study Participants Who Completed Protocol: This analysis includes all study participants who completed the protocol (n = 26)
Arm/Group | All Study Participants Who Completed Protocol
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 71 [58 to 92]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution: male versus female
  Participants
    Female | 5
    Male | 21
Region of Enrollment [Number; unit: participants] — Regions of subject enrollment
  participants
    United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Visit 1 Until Visit 2) to Endpoint (After Visit 2 Until Visit 3) in the Freezing of Gait Questionnaire Score.
Description: The FOGQ has a minimum of 0 and max of 4 for each question, with 4 representing more severe freezing of gait. There are 6 questions, so the total score ranges from 0 to 24. It was pre-specified that all 26 subjects were treated as a single group with respect to the primary outcome measure regardless of whether or not they had a 1 month or 2 month baseline period.
Time Frame: 2-3 months
Population: These 13 subjects were those who were reandomized to a 1 month baseline before use of the laserlight visual cue.
Measure: Mean (Standard Error); unit: change in FOGQ score
Groups:
- 1 Month Baseline Before Use of Laserlight Visual Cue: subjects had a 1 month baseline before use of laserlight visual cue
Arm/Group | 1 Month Baseline Before Use of Laserlight Visual Cue
Number analyzed (Participants) | 13
change in FOGQ score | 1.25 (0.48)
Statistical Analysis 1: Comparison: 1 Month Baseline Before Use of Laserlight Visual Cue; Test type: Superiority; p = 0.0152, t-test, 2 sided; two-tailed paired t-test; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [0.26 to 2.23], Standard Error of Mean 0.48

2. Secondary Outcome: Mean Change in Time to Perform the Timed Gait Test With vs Without the Laser Feature
Description: Mean change in time to perform the timed gait test with versus without the laser feature from visit 1 to visit 3. It was pre-specified that all 26 subjects would be treated as a single group with respect to the outcome measure regardless of whether or not they had a 1 month or 2 month baseline period
Time Frame: 2-3 months
Population: All 26 subjects who entered the study and completed the protocol, so this excludes the 6 subjects who dropped out before any exposure to the laserlight visual cue
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- All Study Participants Who Completed Protocol: All 26 subjects who entered the study and completed the study protocol.
Arm/Group | All Study Participants Who Completed Protocol
Number analyzed (Participants) | 26
seconds
  Before laserlingh visual cue | 65 (26.2)
  With the laserlight visual cue | 57.6 (23.3)
Statistical Analysis 1: Comparison: All Study Participants Who Completed Protocol; Test type: Superiority; p = 0.005, t-test, 2 sided; Mean Difference (Final Values) = 50, 95% CI 2-sided [23.9 to 76.1], Standard Error of Mean 11.7

3. Secondary Outcome: Mean Change in Number of Falls Without Versus With the Laserlight Visual Cue.
Description: Mean change in falls per week for the period between visit 1 and visit 2 (without laserlight visual cue) compared to the period between visit 2 and visit 3 (with the laserlight visual cue).
Time Frame: 2-3 months
Population: 10 Study Participants who completed protocol and who met a predetermined criterion for this subgroup analysis by experiencing one or more falls during both baseline and the subsequent study period. This excludes the 6 subjects who dropped out before any exposure to the laserlight visual cue
Measure: Mean (Standard Deviation); unit: falls per week
Groups:
- All Study Participants Who Completed Protocol: All 26 Study Participants who completed protocol. This excludes the 6 subjects who dropped out before any exposure to the laserlight visual cue.
Arm/Group | All Study Participants Who Completed Protocol
Number analyzed (Participants) | 10
falls per week
  without laserlight visual cue | 3.23 (1.31)
  with laserlight visual cue | 2.12 (0.92)
Statistical Analysis 1: Comparison: All Study Participants Who Completed Protocol; two-tailed Wilcoxan signed-rank sum test; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney); two-tailed Wilcoxan signed-rank sum test; Mean Difference (Net) = 1.11, Standard Deviation 1.31

4. Secondary Outcome: Percentage Change in Falls
Description: The mean change in fall frequency from the baseline period without the laserlight visual cue compared to the subsequent period during which they used the laserlight visual cue among subjects experiencing at least one fall during the baseline and subsequent study periods. This outcome measure is expressed as a percentage change from the baseline period.
Time Frame: 1 to 2 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % change in fall frequency
Groups:
- 1 or 2 Month Baseline Before Use of Laserlight Visual Cue: subjects had a 1 month baseline before use of laserlight visual cue
Arm/Group | 1 or 2 Month Baseline Before Use of Laserlight Visual Cue
Number analyzed (Participants) | 10
% change in fall frequency | 39.5 (9.3)
Statistical Analysis 1: Comparison: 1 or 2 Month Baseline Before Use of Laserlight Visual Cue; The percentage change in falls was analyzed using a two-tailed one-sample t-test with a hypothesized mean of 0; Test type: Other — The percentage change in falls was analyzed using a two-tailed one-sample t-test with a hypothesized mean of 0; p = 0.002, t-test, 2 sided — Two-tailed one-sample t-test with a hypothesized mean of 0. This analysis was not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: Average of 6.5 weeks per subject
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No